CLINICAL TRIAL: NCT05140057
Title: Preparation Regimens to Improve Capsule Endoscopy Visualization and Diagnostic Yield: a Randomized Trial
Brief Title: Preparation Regimens to Improve Capsule Endoscopy Visualization and Diagnostic Yield
Acronym: PrepRICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Responsible Party: Principal Investigator, Maria Manuela Estevinho, Medical Doctor, Principal Investigator, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0001
Record Dates: First submitted 2021-10-05; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Obscure Gastrointestinal Bleeding
Keywords: Small bowel capsule endoscopy; Obscure gastrointestinal bleeding; Bowel preparation
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Protocol 1 (Experimental): 1L of Moviprep® solution the night before the procedure
  Interventions: Combination Product: Moviprep
- Protocol 2 (Experimental): 1L of Moviprep® solution up to 2h before the procedure
  Interventions: Combination Product: Moviprep
- Protocol 3 (Experimental): 0.5L of Moviprep® solution up to 2h before the procedure plus 0.5L of Moviprep® solution after the capsule had reached the duodenum
  Interventions: Combination Product: Moviprep
- Protocol 4 (Experimental): 1L of Moviprep® solution after the capsule had reached the duodenum
  Interventions: Combination Product: Moviprep

INTERVENTIONS:
Combination Product: Moviprep — Bowel preparation for small bowel capsule endoscopy - same product for all groups, different administration timings

SUMMARY:
Small bowel capsule endoscopy (SBCE) has become an important tool in clinical practice since its introduction in 2000. This non-invasive method allows the visualization of small bowel mucosa, being essential in the management of many conditions, such as suspected small bowel bleeding, inflammatory bowel diseases and intestinal polyposis syndromes. Despite recommendations concerning SBCE in different pathologies, there are still some technical concerns to be addressed. The optimal preparation for SBCE has been one of these controversial issues.

Currently, the European Society of Gastrointestinal Endoscopy (ESGE) recommends that patients ingest a purgative agent (2L of polyethylene glycol, PEG) and antifoaming agents for SBCE, because it was associated with a better visualization. However, it remains unclear which is the optimal timing for purgative use. Furthermore, the use of a booster agent after capsule ingestion is already performed in colon capsule endoscopy, but less is known about its application in SBCE. Also, it remains to be clarified whether a better visualization results in higher diagnostic yield and impacts patients' outcomes.

Therefore, the global aim of this prospective, randomized, multi-centric study is to determine the optimal timing and preparation for small-bowel capsule endoscopy (regardless of the equipment used), comparing four groups of different preparation protocols:

* Protocol 1) 1L of Moviprep® solution the night before the procedure
* Protocol 2) 1L of Moviprep® solution up to 2h before the procedure
* Protocol 3) 0.5L of Moviprep® solution up to 2h before the procedure plus 0.5L of Moviprep® solution after the capsule had reached the duodenum (assessed with real-time viewer)
* Protocol 4) 1L of Moviprep® solution after the capsule had reached the duodenum (assessed using real-time viewer)

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or older
* Present OGIB (either occult or overt)
* Agree with study's procedures and have signed the informed consent for the study and SBCE, prior to SBCE procedure

Exclusion Criteria:

* Patients performing capsule endoscopy in urgent setting for overt obscure GI bleeding
* Inpatients or bedridden
* History of surgery of the esophagus, stomach, small bowel, or colon
* History of abdominal or pelvic radiation therapy
* Suspected or confirmed stenosis or occlusion
* Suspected or confirmed bowel perforation
* Severe comorbidities, as defined by grade 3 "severe decompensation" in the Adult Comorbidity Evaluation-27 index (ACE-27)
* Pregnant women
* Patients using narcotics or prokinetics in the week before the SBCE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | During the procedure
  Proportion of SBCE with positive findings. findings will be classified based on the Saurin classification; the investigators will consider a positive SBCE when lesions classified as P2 or active bleeding are detected (Saurin classification, Table 2), the remaining will be classified as negative
Adequate cleansing rate | During the procedure
  A cutoff value of quantitative index ≥ 8 points

SECONDARY OUTCOMES:
Proportion of SBCE with vascular lesions | During the procedure
  Vascular lesions identified in each tertile
Proportion of SBCE with active bleeding | During the procedure
  Active bleeding in each tertile
Diagnostic yield per tertile | During the procedure
  Positive findings in each tertile
Transit times | During the procedure
  Time of entry in the stomach, duodenum and cecum
Symptoms experienced during SBCE procedure | During the procedure
  Nausea, vomit, bloating, abdominal pain
Overall patients' satisfaction with the cleansing regimen | During the procedure
  rated on a 5-point scale: 1 - very easy, 2 - easy, 3 - intermediate, 4 - difficult, 5 - very difficult
Small bowel cleansing | During the procedure
  Mean quantitative index of the distal third of small bowel

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No